CLINICAL TRIAL: NCT03874624
Title: Normal Values for Myocardial Left Atrial Strain
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Fundació Institut de Recerca de l'Hospital de la Santa Creu i Sant Pau (Other)
Responsible Party: Sponsor
Other Study IDs: IIBSP-STR-2018-111
Record Dates: First submitted 2019-03-01; First posted 2019-03-14 (Actual); Last update posted 2019-03-14 (Actual); Status verified 2019-03

CONDITIONS: Atrial Function

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Diagnostic Test: two-dimensional speckle tracking — Analysis of myocardial left atrial strain using two-dimensional speckle tracking echocardiography.

SUMMARY:
Transversal retrospective and unicentric study. The investigators sought to determine the normal values for two-dimensional myocardial left atrial strain for the cardiology ultrasound system available in their centre (Philips EPIQ ultrasound machine and 10.8.5 QLAB cardiac analysis software). Studies performed in their department which meet the criteria for an adequate strain analysis will be retrospectively reviewed.

ELIGIBILITY:
Inclusion Criteria:

* No history of cardiopathy / pneumopathy.
* No history of hypertension or mellitus diabetes.

Exclusion Criteria:

* Pregnancy.
* Athletes.
* Body mass index < 16 or => 30 kg/m2.
* Previous treatment with cardiotoxic chemotherapy.
* Dilated left ventricle (telediastolic diameter index > 30 mm/m2).
* Interventricular septal thickness => 12 mm.
* Dilated left atria (volume => 31 ml/m2).
* Systolic pulmonary pressure => 35 mmHg.
* Moderate or severe valvulopathy.
* Incomplete or suboptimal left atrial visualization.
* Frame rate < 50 fps.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Healthy controls.
Sampling Method: Non-Probability Sample
Enrollment: 43 (Estimated)
Dates: Start 2019-02-22 (Actual); Primary Completion 2019-05-31 (Estimated); Study Completion 2019-05-31 (Estimated)

PRIMARY OUTCOMES:
Global peak reservoir strain. | Through study completion, an average of 4 months.
  Percentage of peak reservoir strain for 4-, 2- and 3-chambers will be combined to report percentage of global peak reservoir strain.
Global pump strain. | Through study completion, an average of 4 months.
  Percentage of pump reservoir strain for 4-, 2- and 3-chambers will be combined to report percentage of global pump strain.
Global conductance strain. | Through study completion, an average of 4 months.
  Measured as the difference between global reservoir strain and gobal pump strain.
Global reservoir strain rate. | Through study completion, an average of 4 months.
  Reservoir strain rate for 4-, 2- and 3-chambers will be combined to report global reservoir strain rate.
Global conductance strain rate. | Through study completion, an average of 4 months.
  Conductance strain rate for 4-, 2- and 3-chambers will be combined to report global conductance strain rate.
Global pump strain rate. | Through study completion, an average of 4 months.
  Pump strain rate for 4-, 2- and 3-chambers will be combined to report global pump strain rate.

SECONDARY OUTCOMES:
Age in years | Through study completion, an average of 4 months.
Sex | Through study completion, an average of 4 months.
  male or female
Weight in kilograms | Through study completion, an average of 4 months.
Height in meters | Through study completion, an average of 4 months.
Left atrial volume | Through study completion, an average of 4 months.
  Measured by biplanar volumetric method
Left ventricular ejection fraction | Through study completion, an average of 4 months.
  Measured by biplanar Simpson's method
Left ventricular telediastolic volume | Through study completion, an average of 4 months.
  Measured by Simpson's method
Left ventricular dimensions | Through study completion, an average of 4 months.
  Assessed by the following parameters: telediastolic diameter, interventricular septal thickness, posterior wall thickness (in mm)
E/A ratio | Through study completion, an average of 4 months.
  Transmitral flow profile.
E/e' ratio | Through study completion, an average of 4 months.
  Tissue doppler derived parameter.

CONTACTS AND LOCATIONS:
Locations (1):
- Hospital de la Santa Creu i Sant Pau, Barcelona, Spain